CLINICAL TRIAL: NCT04905615
Title: The Use of Data From Wearable Technology to Co-develop School-specific Physical Activity Interventions in Children Aged 9-11
Brief Title: The Use of Data From Wearable Technology to Co-develop School-specific Physical Activity Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other); University of Bristol (Other); Loughborough University (Other)
Responsible Party: Principal Investigator, Georgina Wort, Principal Investigator, University of Bath
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: EP 1920 009
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Physical Activity
Keywords: Physical Activity; Primary School Children; Wearable Technology; Data Driven Intervention; School-based Intervention; Co-design
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Measures (No Intervention): The first two-weeks within each school children's baseline physical activity data will be collected. Children will be blinded to the data, receiving no feedback. Teachers will be instructed not to change normal school practices or encourage children's physical activity.
- Data-Driven Strategy Based Intervention (Experimental): During the following 2-weeks teachers will be implementing strategies to improve their class' physical activity. These are individualised strategies which will be co-developed during semi-structured interviews where teachers will discuss data visualisations with the researcher which depicts their class' physical activity over the 2-week baseline period. Teachers will then implement these strategies over the subsequent 2-weeks. During this time teachers are able to share the physical activity data with their pupils if they wish.
  Interventions: Other: Data-driven and teacher led school based strategies.

INTERVENTIONS:
Other: Data-driven and teacher led school based strategies. — The intervention is individualised to each school, depending on the teacher led strategies which are data-informed
  Arms: Data-Driven Strategy Based Intervention

SUMMARY:
Increasing physical activity is vital for children's physical and mental health. It is important to address inactivity early and engage children in positive behaviours which can be sustained throughout life. Teachers are well placed to understand and influence in-school factors impacting children's physical activity. As wearable technologies continue to improve and become more accessible, they offer the opportunity to engage schools in the data collection process, as well as providing them with the capacity to monitor strategies designed to improve physical activity. This study is a within-subject, pre-post, co-developed intervention design.

DETAILED DESCRIPTION:
Previous interventions have not successfully increased physical activity levels in primary schools. This is arguably due to a lack of comprehensive data collection methods and the lack of co-involvement of teachers and children in intervention design. In previous research, accelerometers have been used by researchers to quantify children's physical activity levels. However, these have been research-grade devices which require a more complex analysis to extract results; because of this, these types of measurement tools have not been utilised by schools. This study will aim to utilise user-friendly technologies which can engage schools in the data collection process and be employed by schools to implement and measure strategies designed to increase physical activity by providing immediate feedback.

This project aims to investigate whether data from wearable technologies can be used to inform primary school-based practices and improve children's physical activity within school hours using co-developed interventions. This project is a participatory mixed-methods design in two phases. 7-9 schools will be recruited. The first phase in each school involves baseline measures of pupils' physical activity for 2-weeks, using accelerometers which have been specifically designed for school use. Pupils will be blinded to the physical activity data during this period. During this 2-week baseline teachers will be instructed to carry out lessons as normal, not changing their behaviour, or encouraging the pupils' physical activity. Data visualisations will be created from the 2-weeks of physical activity data collected within each school. Teachers will then be interviewed online, using Microsoft Teams, and encouraged to reflect on the physical activity data and co-develop 3-5 action points or strategies to increase children's physical activity. Teachers will then be asked to implement these action points over the subsequent 2-weeks, where again children's physical activity will be measured with the accelerometers. This time children will not be blinded to the data and can receive physical activity feedback if this is a strategy selected by their teacher. These changes will be at each schoolteacher's discretion and managed in a way they deem most appropriate. Following these 2-week changes teachers will be interviewed again about their experiences of using the technology and implementing strategies to encourage physical activity. They will then be shown similar data visualisations as before, comparing changes in pupils' physical activity between each 2-week period.

ELIGIBILITY:
Inclusion Criteria:

* Any pupil from the each respective UK-based school and class. Pupils in years 5 to 6 (aged 9-11 years old).

Exclusion Criteria:

* No exclusion criteria.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Teachers input the gender pupils identify with into the physical activity data collection software.
Enrollment: 228 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Step Count | 2-weeks baseline, compared to 2-weeks intervention period in each school
  Changes in step counts from baseline

SECONDARY OUTCOMES:
Moderate to Vigorous Physical Activity (MVPA) | 2-weeks baseline, compared to 2-weeks intervention period in each school
  Changes in MVPA from baseline
Qualitative Data | Interviews conducted at the end of each 2-week period with each class teacher.
  The first interview with teachers is conducted following the 2-week baseline measures, during which their class' physical activity data will be discussed and action points co-developed. The second interview will take place after the 2-week intervention period. Teachers will be presented with their class' physical activity data changes, which will be discussed alongside the successes and challenges of the implemented action points.
Pupil Demographics and Physical Activity Measures | 4 weeks
  Physical activity changes in different demographic groups (i.e., gender, free school meal, pupil premium and SEN)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Banes, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided